CLINICAL TRIAL: NCT05950997
Title: A Single Arm Study of Acalabrutinib Combined With Obinutuzumab in Chinese Patients With Treatment-Naive Chronic Lymphocytic Leukemia
Brief Title: A Single Arm Study of Acalabrutinib Conbimed With Obinutuzumab in Chinese Patients With Previously Untreated CLL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-22-22033
Record Dates: First submitted 2023-06-15; First posted 2023-07-18 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; obinutuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- previously untreated chronic lymphocytic leukemia. (Experimental): Previously untreated CLL patients with ≥1 of the IWCLL 2018 criteria for requiring treatment will be enrolled. Treatment with acalabrutinib may be continued until treatment for 24 months, or until an unacceptable drug-related toxicity occurs or until disease progression, whichever occurs first. Dose modification provisions are provided in the study protocol. Treatment with obinutuzumab or obinutuzumab/chlorambucil is up to 6 cycles per the obinutuzumab package insert.
  Interventions: Drug: Acalabrutinib; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Acalabrutinib — 100 mg capsules administered by mouth once daily (28-day cycles)
Drug: Obinutuzumab — 100 mg administered intravenously on Day 1 and 900 mg administered intravenously on Day 2, 1000 mg administered intravenously on Day 8 and 15 of cycle 2 and 1000 mg on Day 1 of subsequent cycles for a total of 6 cycles (28-day cycles)

SUMMARY:
This is a single-arm, prospective study to assess the efficacy and safety of acalabrutinib combined with obinutuzumab in subjects with previously untreated chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
Subject participation will include a Screening Phase, a Treatment Phase, a Follow-up Phase.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥18 years of age.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 with no deterioration over the previous 2 weeks prior to baseline or day of first dosing
3. Diagnosis of CD20+ CLL that meets published diagnostic criteria(Hallek 2018):

   1. Monoclonal B cells (either kappa or lambda light chain restricted) that are clonally co-expressing ≥ 1 B-cell marker (CD19, CD20, or CD23) and CD5.
   2. Prolymphocytes may comprise ≤ 55% of blood lymphocytes.
   3. Presence of ≥ 5 x 109 B lymphocytes/L (5000 μL) in the peripheral blood (at any point since diagnosis).
4. Active disease meeting ≥ 1 of the following iwCLL 2018 criteria for requiring treatment:

   1. Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia (hemoglobin < 10 g/dL) and/or thrombocytopenia (platelets < 100,000/μL).
   2. Massive (i.e., ≥ 6 cm below the left costal margin), progressive, or symptomatic splenomegaly.
   3. Massive nodes (i.e., ≥ 10 cm in the longest diameter), progressive, or symptomatic lymphadenopathy.
   4. Progressive lymphocytosis with an increase of > 50% over a 2-month period or (lymphocyte doubling time) LDT of < 6 months. LDT may be obtained by linear regression extrapolation of ALC obtained at intervals of 2 weeks over an observation period of 2 to 3 months. In subjects with initial blood lymphocyte counts of < 30 x 109/L (30,000/μL) may require a longer observation period to determine the LDT. In addition, factors contributing to lymphocytosis or lymphadenopathy other than CLL (e.g., infections) should be excluded.
   5. Autoimmune anemia and/or thrombocytopenia that is poorly responsive to corticosteroids.
   6. Constitutional symptoms documented in the subject's chart with supportive objective measures, as appropriate, defined as ≥ 1 of the following disease-related symptoms or signs:

   i Unintentional weight loss ≥ 10% within the previous 6 months before Screening.

   ii Significant fatigue (i.e., ECOG performance status 2; inability to work or perform usual activities).

   iii Fevers higher than 100.5°F or 38.0°C for 2 or more weeks before Screening without evidence of infection.

   iv Night sweats for > 1 month before Screening without evidence of infection.
5. Meet the following laboratory parameters:

   1. ANC ≥ 750 cells/μL (0.75 x 109/L), or ≥ 500 cells/μL (0.50 x 109/L) in subjects with documented bone marrow involvement, and independent of growth factor support 7 days before assessment.
   2. Platelet count ≥ 50,000 cells/μL (50 x 109/L), or ≥ 30,000 cells/μL (30 x 109/L) in subjects with documented bone marrow involvement, and without transfusion support 7 days before assessment. Subjects with transfusion-dependent thrombocytopenia are excluded.
   3. Serum AST and ALT ≤3 x upper limit of normal (ULN).
   4. Total bilirubin ≤1.5 x ULN, unless directly attributable to Gilbert's syndrome
   5. Estimated creatinine clearance of ≥30 mL/min, calculated by Cockcroft-Gault (using actual body weight), or serum creatinine ≤2×ULN, (if male, [140-Age] x Mass [kg] / [72 x creatinine mg/dL]; multiply by 0.85 if female)
6. Female subjects who are sexually active and can bear children must agree to use highly effective forms of contraception while on the study and for 2 days after the last dose of acalabrutinib, or 18 months after the last dose of obinutuzumab, whichever is longer.
7. Male subjects who are sexually active must agree to use highly effective forms of contraception with the addition of a barrier method (condom) during the study and for 90 days after the last dose of Obinutuzumab, whichever is later.
8. Men must agree to refrain from sperm donation during the study and for 90 days after the last dose of Obinutuzumab, whichever is later.
9. Willing and able to participate in all required evaluations and procedures in this study protocol, including swallowing capsules and tablets without difficulty.
10. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local patient privacy regulations).

Exclusion Criteria:

1. Evidence of disease (such as severe or uncontrolled systemic diseases, including uncontrolled hypertension and renal transplant) that, in the investigator's opinion, make it undesirable for the patient to participate in the study or that would jeopardize compliance with the protocol.
2. Any prior systemic treatment for CLL (note: Prior localized radiotherapy is allowed).
3. Known CNS lymphoma or leukemia.
4. Known prolymphocytic leukemia or history of, or currently suspected, Richter's syndrome.
5. Uncontrolled AIHA or ITP defined as declining hemoglobin or platelet count secondary to autoimmune destruction within the screening period or requirement for high doses of steroids (> 20 mg daily of prednisone daily or equivalent).
6. Corticosteroid use > 20 mg within 1 week before first dose of study drug, except as indicated for other medical conditions such as inhaled steroid for asthma, topical steroid use, or as premedication for administration of study drug or contrast. For example, subjects requiring steroids at daily doses > 20 mg prednisone equivalent systemic exposure daily, or those who are administered steroids for leukemia control or WBC count lowering are excluded.
7. Major surgery within 30 days before first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
8. History of prior malignancy that could affect compliance with the protocol or interpretation of results, except for the following:

   1. a. Curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or carcinoma in situ of the prostate at any time prior to study.
   2. b. Other cancers not specified above that have been curatively treated by surgery and/or radiation therapy from which subject is disease-free for ≥3 years without further treatment.
9. Significant cardiovascular disease such as symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification at Screening. Note: Subjects with controlled, asymptomatic atrial fibrillation are allowed to enroll on study.
10. History of or ongoing confirmed progressive multifocal leukoencephalopathy (PML).
11. Received any investigational drug within 30 days or 5 half-lives (whichever is shorter) before first dose of study drug.
12. Refractory nausea and vomiting, inability to swallow the formulated product, or malabsorption syndrome; chronic gastrointestinal disease, gastric restrictions, or bariatric surgery such as gastric bypass; partial or complete bowel obstruction, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of study treatment.
13. Received a live virus vaccination within 28 days of first dose of study drug.
14. Known history of infection with HIV.
15. Any active significant infection (e.g., bacterial, viral or fungal, including subjects with positive cytomegalovirus [CMV] DNA polymerase chain reaction [PCR]).
16. Serologic status reflecting active hepatitis B or C infection.

    1. Subjects who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antigen (HBsAg) negative will need to have a negative PCR result before randomization and must be willing to undergo DNA PCR testing during the study. Those who are HbsAg-positive or hepatitis B PCR positive will be excluded.
    2. Subjects who are hepatitis C antibody positive will need to have a negative PCR result before randomization. Those who are hepatitis C PCR positive will be excluded.
17. History of stroke or intracranial hemorrhage within 6 months before first dose of study drug.
18. History of bleeding diathesis (e.g., hemophilia, von Willebrand disease).
19. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists.
20. Requires treatment with a strong cytochrome P450 3A (CYP3A) inhibitor or inducer. The use of strong CYP3A inhibitors within 1 week or strong CYP3A inducers within 3 weeks of the first dose of study drug is prohibited.
21. Breastfeeding or pregnant.
22. Concurrent participation in another therapeutic clinical trial.
23. Requires treatment with proton-pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole).
24. Current life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the subject's safety or put the study at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate at 24 months | At 24 months
  24-month progression-free survival rate is defined as the proportion of subjects without progression or death due to any cause at 24 months since the start of study drug. The evaluation of progression will be investigator-assessed per International Workshop on Chronic Lymphocytic Leukemia criteria(iwCLL2018) criteria.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 24 months after LPI
  ORR is defined as the proportionof subjects with complete remission (CR), complete remission with incomplete bone marrow recovery (CRi), nodular partial remission(nPR), or partial remission(PR) assessed by investigator per iwCLL2018 criteria.
Duration of response (DOR) | At 24 months
  DOR is defined as the time from the first documentation of objective response to the earlier time of disease progression (assessed by the investigator, per iwCLL 2018 criteria) or death from any cause. The same censoring rules and analysis methods will be applied as described for PFS.
24-month overall survival rate (24m OS rate) | At 24 months
  24-month overall survival rate is defined as the proportion of subjects without death due to any cause at 24 months since the start of study drug.
Adverse Events (AEs) | Up to acalabrutinib treatment for 24 months
  AEs will be graded by the investigator according the NCI CTCAE v5.0 or higher for hematologic and nonhematologic AEs. Each AE verbatim term will be coded to a system organ class and a preferred term using the Medical Dictionary for Regulatory Activities (MedDRA).
Treatment-Emergent Adverse Events | Up to acalabrutinib treatment for 24 months
  All treatment-emergent adverse events (TEAEs) will be summarized. In addition, AE incidence rates will also be summarized by severity and relationship to study drug.
  Grade 3 or Grade 4 TEAEs; TEAEs leading to permanent study drug treatment discontinuation; TEAEs leading to dose reduction; serious TEAEs; and TEAEs resulting in death will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Jianyong Li, PhD, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Department of Haematology, the First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital, Nanjin, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No